CLINICAL TRIAL: NCT02304796
Title: Randomized Controlled Trial Examining the Effectiveness of Two Group Psychotherapies for Anxiety Disorders: Unified Cognitive-behavioral Therapy vs. Combined Cognitive Behavioral and Dance/Movement Therapy
Brief Title: Unified Cognitive-Behavioral Therapy (CBT) vs. Combined CBT and Dance/Movement Therapy (DMT) for Anxiety Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0015-14-SHA
Record Dates: First submitted 2014-11-22; First posted 2014-12-02 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Anxiety Disorders
Keywords: Anxiety Disorders; Group Psychotherapy; Cognitive-Behavioral Therapy; Dance/Movement Therapy; CBT; DMT; Unified Protocol
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unified CBT (Experimental): Group psychotherapy according to the principles of the Cognitive-Behavioral Unified Protocol for Trans-diagnostic Treatment of Emotional Disorders (Barlow et al., 2011).
  Interventions: Behavioral: Unified Cognitive-Behavioral Therapy
- Combined CBT-DMT (Experimental): Group psychotherapy combining cognitive-behavioral principles and techniques with dance/movement therapy techniques.
  Interventions: Behavioral: Combined Cognitive-Behavioral and Dance/Movement Therapy

INTERVENTIONS:
Behavioral: Unified Cognitive-Behavioral Therapy — 20 weekly sessions (1.5-2 hours each), based on the principles of the Unified Protocol for Trans-diagnostic Treatment of Emotional Disorders (Barlow et al., 2011) adapted for a group format.
  The treatment will include 8 different modules of varying length: motivation enhancement, understanding emotions, identifying and monitoring emotions, emotional awareness training, cognitive appraisal and reappraisal, emotional avoidance, emotion driven behaviors, awareness and tolerance of bodily sensations, relapse prevention.
  Arms: Unified CBT
Behavioral: Combined Cognitive-Behavioral and Dance/Movement Therapy — 20 weekly sessions (1.5-2 hours each), based on combined cognitive-behavioral techniques (psychoeducation, awareness and tolerance of emotions, interoceptive exposures, in-vivo exposures, cognitive flexibility) and dance/movement techniques.
  Arms: Combined CBT-DMT

SUMMARY:
The current pilot study will examine and compare the effectiveness of two group psychotherapies for mixed anxiety disorders: 1. unified cognitive-behavioral protocol, adapted to a group format. 2. combined cognitive-behavioral and dance/movement therapy.

In addition, change in proposed mechanism in each therapy will be examined, along with their association with change in outcome measures during therapy.

DETAILED DESCRIPTION:
The current pilot study will examine and compare the effectiveness of two group psychotherapies for mixed anxiety disorders: 1. unified cognitive-behavioral protocol, adapted to a group format. 2. combined cognitive-behavioral and dance/movement therapy.

24 patients will be randomized to 1 of the two treatment arms and treated with 20 weekly 1.5-2 hours therapy sessions. Independent evaluator and self-reports measures will be collected at intake, pre-treatment, session by session, post-treatment and and follow-up.

Hypotheses:

1. Both groups will show effectiveness, as revealed by reduction in anxiety severity and increase in valued living.
2. Changes in process measures (proposed mechanism of change - emotion regulation, working alliance, fear of bodily sensations, bodily/movement awareness) will be predictive of change in outcome measures (anxiety severity and valued living).
3. Changes in bodily/movement awareness will be more predictive of change in outcome measures in the CBT-DMT group than in the unified protocol group.

ELIGIBILITY:
Inclusion Criteria:

* One of the following primary axis I DSM-IV-TR diagnoses: Panic disorder with or without Agoraphobia; Social Anxiety Disorder; Generalized Anxiety Disorder; Anxiety Disorder Not Otherwise Specified; Adjustment Disorder With Anxiety; Adjustment Disorder With Mixed Anxiety and Depressed Mood
* If on medication or in other types of treatments, patients must be willing to remain stable on their treatment for the duration of the acute phase of the study (5-6 months)
* Provision of written informed consent

Exclusion Criteria:

* Current or past schizophrenia, psychosis, or bipolar disorder.
* Current suicidal ideation.
* Current substance/alcohol dependence or abuse.
* Cluster A or B personality disorder.
* Pregnancy (for women).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Anxiety Rating Scale | Intake (entry to study), Pre-treatment (1 month from intake), Post-Treatment (6 months from intake), Follow-Up (7 months from intake)
  Structured independent evaluator interview for assessing severity of anxiety

SECONDARY OUTCOMES:
Change in Depression, Anxiety, Stress Scales-21 | Intake (entry to study), Weekly during treatment (weekly between 1-6 months from intake), Post-Treatment (6 months from intake), Follow-Up (7 months from intake)
  Self-report measure of depression, anxiety and stress
Change in Valued Living Questionnaire | Intake (entry to study), Pre-treatment (1 month from intake), Mid-Treatment (3.5 months from intake), Post-Treatment (6 months from intake), Follow-Up (7 months from intake)
  Self-report measure of valued living
Change in Mini International Neuropsychiatric Interview | Intake (entry to study), Pre-treatment (1 month from intake), Post-Treatment (6 months from intake), Follow-Up (7 months from intake)
  Structured independent evaluator interview for assessing Diagnostic and Statistical Manual of Mental Disorders IV Text Revision (DSM-IV-TR) axis I diagnoses

OTHER OUTCOMES:
Change in Difficulties in Emotion Regulation Scale | Intake (entry to study), Weekly during treatment (weekly between 1-6 months from intake), Post-Treatment (6 months from intake), Follow-Up (7 months from intake)
  Self-report measure of different aspects of emotion regulation difficulties
Change in Body Sensations Questionnaire | Intake (entry to study), Pre-treatment (1 month from intake), Mid-Treatment (3.5 months from intake), Post-Treatment (6 months from intake), Follow-Up (7 months from intake)
  Self-report measure of fear of bodily sensations
Change in Bodily Awareness of Emotions Subscale of the Emotion Awareness Questionnaire - Revised | Intake (entry to study), Pre-treatment (1 month from intake), Mid-Treatment (3.5 months from intake), Post-Treatment (6 months from intake), Follow-Up (7 months from intake)
  Self-report measure of awareness of bodily sensations/movement and their emotional meaning
Change in Working Alliance Inventory - Short and Revised form - Group version | Intake (entry to study), Pre-treatment (1 month from intake), Session 5 (2 months from intake), Mid-Treatment (3.5 months from intake), Post-Treatment (6 months from intake), Follow-Up (7 months from intake)
  Self-report measure of working alliance in group therapy

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Bloch, M.D., Principal Investigator — Shalvata Mental Health Center
Locations (1):
- Shalvata Mental Health Center, Hod HaSharon, Israel

REFERENCES:
- [Background] Barlow DH, Farchione TJ, Fairholme CP, Ellard KK, Boisseau CL, Allen LB, Ehrenreich-May J. The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders: Therapist Guide. New York: Oxford University Press: 2011.